CLINICAL TRIAL: NCT03314285
Title: Placebo-Controlled Trial of Evaluation of Sleep Quality in Patients With Chronic Neck Pain
Brief Title: Evaluation of Sleep Quality in Patients With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alper Mengi (Other Government)
Responsible Party: Sponsor-Investigator, Alper Mengi, Physiatrist, Medical Doctor, Gaziosmanpasa Research and Education Hospital
Organization: Gaziosmanpasa Research and Education Hospital (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 04.10.2017/79
Record Dates: First submitted 2017-10-12; First posted 2017-10-19 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Neck Pain; Sleep
Keywords: Cervicalgia
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neck Pain (Other): Patients with chronic mechanical neck pain will be evaluated for sleep quality by the Pittsburgh Sleep Quality Scale.
  Interventions: Other: Sleep Quality
- Healthy volunteers (Other): Healthy volunteers without any disease will be evaluated for sleep quality by the Pittsburgh Sleep Quality Scale.
  Interventions: Other: Sleep Quality

INTERVENTIONS:
Other: Sleep Quality — Sleep quality to be measured by the Pittsburgh Sleep Quality Scale.

SUMMARY:
This study aimed to investigate the effect of chronic neck pain on sleep quality and to determine the factors that may be related to sleep disturbance.

DETAILED DESCRIPTION:
It is thought that chronic neck pain affects sleepiness negatively. However, there are no studies on chronic neck pain and sleep quality. In this study, we would like to determine whether there is a link between chronic neck pain and sleep quality and the factors that may be related.

ELIGIBILITY:
Inclusion Criteria:

* Patient has chronic mechanical neck pain for at least 3 months and without radicular pain
* Patient's visual analogue scale score is 3 and over

Exclusion Criteria:

* History of neurological deficit
* History of cervical stenosis, cervical surgery, spondylolisthesis, scoliosis
* History of central or peripheral nervous system disorders
* History of inflammatory neck pain
* Pregnant or breast feeding
* History of fibromyalgia disease
* History of severe osteoporosis or osteomalacia
* History of infectious, malignancy, and active psychiatric disease
* Noncooperative
* Patient has chronic pain in a region other than the neck region

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2017-11-12 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Pittsburg Sleep Quality Scale | 30 day
  Sleep quality to be measured by the Pittsburgh Sleep Quality Scale.The Pittsburgh Sleep Quality Scale is a 19-item self-rated questionnaire for evaluating subjective sleep quality the previous month. The 19 questions are combined into 7 clinically-derived component scores, each weighted equally from 0-3. The 7 component scores are added to obtain a global score ranging from 0-21, with higher scores indicating worse sleep quality.

SECONDARY OUTCOMES:
Demographic Data | 30 day
  Gender, Age, Education Level, Job
Pain Severity | 7 day
  The pain severity was evaluated using a 10 cm visual analogue scale , where 0 represented no pain, while 10 represented unbearable pain.At evaluation, the average of the pain in activity , in rest , and during the night for the last one week were inquired.

CONTACTS AND LOCATIONS:
Overall Officials: Alper Mengi, M.D., Principal Investigator — Department of Physical Medicine and Rehabilitation, Gaziosmanpasa Taksim Training and Research Hospital
Locations (1):
- Gaziosmanpasa Taksim Research and Education Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No